CLINICAL TRIAL: NCT01643564
Title: Cytokine Profiling of Cardiac Transplant Recipients
Brief Title: Cytokine Profiling Post-Heart Transplant
Status: Terminated | Type: Observational
Why Stopped: Subject Recruitment
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1111M06547
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Transplant
Keywords: Transplant; Cytokines; Graft Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: Heart Transplant Recipients with Unexplained Graft Dysfunction
- Group 2: Normal Control
- Group 3: Class III-IV Heart Failure
- Group 4: Heart Transplant Recipients with Normal Graft Function

SUMMARY:
Measurement of cytokine levels in post-cardiac transplant patients with unexplained graft dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* 18 years and older
* Cardiac Transplant recipient with graft dysfunction of unknown etiology

Group 2

* 18 years or older
* No history of heart failure or cardiac transplantation Group 3
* 18 years or older
* Class II-IV heart failure Group 4
* 18 years or older
* Heart Transplant 6 months or greater prior to blood draw
* No graft dysfunction

Exclusion Criteria:

Group 1 Heart Transplant with Unexplained Graft Dysfunction

* Cellular or antibody-mediated cardiac allograft dysfunction

Group 2 Normal Control group

* Active infection within 1 month of blood draw
* Known Inflammatory Disease

Group 3 Heart Failure Group

* Active infection within 1 month of blood draw
* Known Inflammatory Disease

Group 4 Heart Transplant with Normal Graft Function Group

* Active infection within 1 month of blood draw
* Known graft dysfunction
* Known Inflammatory Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology Clinic and inpatient service. Normal controls are volunteers from within the community.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Differences in cytokine profiles between stable heart transplant recipients and those with acute rejection | 12 months
  Differences in cytokine profiles between stable heart transplant recipients and those with acute rejection

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Eckman, MD, Principal Investigator — University of Minnesota